CLINICAL TRIAL: NCT06902714
Title: Evaluating the Effects of Oral Tranexamic Acid on Short Term Postoperative Outcomes Following Total Shoulder Arthroplasty: A Randomized Control Trial
Brief Title: Effects of Oral Tranexamic Acid on Short Term Postoperative Outcomes Following Total Shoulder Arthroplasty
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Walter Smith, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-300014204; UAB (Other: UAB)
Record Dates: First submitted 2025-03-18; First posted 2025-03-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Shoulder Arthroplasty
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- oral tranexamic acid (Experimental)
  Interventions: Drug: oral tranexamic acid
- Oral Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: oral tranexamic acid — one group of subjects will receive oral tranexamic acid and the other will receive oral placebo
  Arms: oral tranexamic acid
Drug: Placebo — one group of randomized subjects will receive placebo and the other will receive oral tranexamic acid
  Arms: Oral Placebo

SUMMARY:
The purpose of this clinical trial is to evaluate the short-term clinical outcomes of patients undergoing total shoulder arthroplasty who receive an extended postoperative course of oral tranexamic acid

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients (ages 18-79) undergoing primary total shoulder arthroplasty

Exclusion Criteria:

* Patients with Cancer, venous thromboembolism, stroke, heart disease, pregnant or nursing, allergic to TXA, current tobacco use, anticoagulants other than aspirin.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
VAS | 2 weeks
  visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Walter Smith, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States